CLINICAL TRIAL: NCT05905445
Title: The Effect of Ozone Gel as an Adjunct Treatment in Patients of Periodontitis According to Clinical and Biological Marker. A Split-mouth Randomized Controlled Clinical Trial.
Brief Title: Use of Ozone Gel as an Antimicrobial in Treatment of Periodontitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ghufran Falih Hassan (Other)
Responsible Party: Sponsor-Investigator, Ghufran Falih Hassan, postgraduate student, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ozone gel in periodontitis
Record Dates: First submitted 2023-05-26; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Periodontal Pocket; Periodontitis
MeSH Terms: conditions — Periodontal Pocket; Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ozone gel with conventional scaling and root planning (Experimental): administered ozone gel in the probing pocket depth after scaling and root planning by a disposable plastic syringe with a blunt tip until the access ozone became out of the pocket. this procedure is made at baseline and in the first month. instructed the patient not to eat or drink for at least 30 minutes
  Interventions: Drug: ozone gel
- only conventional scaling and root planning (No Intervention): only scaling and root planning without any intervention.

INTERVENTIONS:
Drug: ozone gel — the activity of omega-3 in the ozone gel may be advantageous as a host-modulating agent in the supplemental treatment of periodontitis
  Arms: ozone gel with conventional scaling and root planning

SUMMARY:
Periodontitis is an inflammatory disease that destroys tooth-supporting structures through oral bacterial plaque. ozone gel's act as an antimicrobial effect as an adjunct to conventional periodontal therapy (scaling and root planning). exposure of bacteria to ozone leads to the oxidation of the phospholipids and lipoproteins that comprise the bacterial cell membrane. Ozone gel has the potential to play an anti-inflammatory role in the treatment of periodontitis by monitoring both clinical and biological parameters.

DETAILED DESCRIPTION:
Periodontitis is an inflammatory disease that destroys tooth-supporting structures through oral bacterial plaque. Scaling and root planning are considered the gold standard treatment for periodontal disease. Antiseptics represent an aid to the gold standard nonsurgical treatment of scaling and root planning (SRP) for periodontal disease. Adjuncts to scaling and root planning have been introduced as ozone gel. This gel represents both antimicrobial and beneficial effects while expressing safe cytocompatibility toward host tissues, which is progressively developing.

The study aims to determine ozone gel's antimicrobial effect as an adjunct to conventional periodontal therapy (scaling and root planning).

Material and Methods: Twenty-one patients with periodontitis were enrolled in this study. There were 58 periodontal pockets divided into two groups by a blinded split-mouth design. The control group had 28 periodontal pockets treated with scaling and root planning only, while the test group had 30 with scaling and root planning and ozone gel. Two gel applications were applied at baseline and one month after the treatment. Plaque index, bleeding on probing, probing pocket depth, and relative attachment level were recorded. Gingival crevicular fluid samples were collected from the pockets at each site for both groups at different time intervals. The GCF sample was transferred into Eppendorf tubes containing 1.5 ml of PBS buffer, and the samples were stored in a freezer at -40˚C.

ELIGIBILITY:
Inclusion Criteria:

* The patient should be systemically healthy
* The patient has periodontitis equal to or more than two non-adjacent teeth, with probing pocket depth equal to or more than 4mm.
* Patients capable of following orders and motivation

Exclusion Criteria:

* Patients with removable dentures who undergo orthodontic therapy.
* Patients with teeth suffer from endo-periodontal lesions.
* Patients have three months of using anti-inflammatory medications, antibiotics, immune suppressants, or oral contraceptives.
* Patients having systemic conditions that affect the condition.
* Pregnant or nursing mothers.
* Patients who are smokers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
probing pocket depth | baseline to one and three months
  change of probing pocket depth by ozone gel as an adjunct to non-surgical treatment

SECONDARY OUTCOMES:
plaque index | baseline to one and three months
  change in presence plaque (used disclosing agent) by ozone gel as an adjunct to non-surgical treatment
bleeding on probing | baseline to one and three months
  change in presence bleeding on probing (used UNC 15 probe) by ozone gel as an adjunct to non-surgical treatment
clinical attachment loss | baseline to one and three months
  change in presence clinical attachment loss (Used relative attachment stent) by ozone gel as an adjunct to non-surgical treatment
level of platelet-activating factor in gingival crevicular fluid | baseline to one and three months
  change in level of platelet-activating factor in gingival crevicular fluid (Used ELISA kit to measurement level of PAF in gingival crevicular fluid) by ozone gel as an adjunct to non-surgical treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ghufran Falih Hassen, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colombo M, Gallo S, Garofoli A, Poggio C, Arciola CR, Scribante A. Ozone Gel in Chronic Periodontal Disease: A Randomized Clinical Trial on the Anti-Inflammatory Effects of Ozone Application. Biology (Basel). 2021 Jul 6;10(7):625. doi: 10.3390/biology10070625. PMID 34356480